CLINICAL TRIAL: NCT00087503
Title: A Phase II Efficacy And Safety Study Intravenous Edotecarin In Patients With Advanced Gastric Cancer That Has Progressed Or Recurred After Prior Fluropyrimidine-Based Chemotherapy
Brief Title: Intravenous Edotecarin in Patients With Advanced Gastric Cancer That Has Progressed or Recurred After Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDOAGA-6736-001; A5921008
Record Dates: First submitted 2004-07-09; First posted 2004-07-13 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — edotecarin

INTERVENTIONS:
Drug: Edotecarin

SUMMARY:
This will be an international, multicenter, uncontrolled, 2-stage, phase II study in adult patients with advanced gastric cancer, reasonable performance status, good organ function, lack of serious concomitant medical conditions. Patients must have progressed or recurred after a fluoropyrimidine-containing regimen at anytime for primary metastatic disease or within 6 months of last dose of adjuvant therapy. Twenty-one evaluable patients will be enrolled in Stage 1. If at least 2 objective tumor responses are observed in the first 21 evaluable patients, the study will be expanded to enroll a total of 41 evaluable patients. Edotecarin will be administered at a starting dose of 13 mg/m2 as an IV infusion over 60 minutes in repeated 3-week cycles treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction adenocarcinoma (i.e., an adenocarcinoma with >50% extension in the stomach)
* Presence of locally advanced or metastatic disease non-amenable to surgery +/- chemo-radiation with curative intent
* Progression or recurrence after a fluoropyrimidine-containing regimen at any time for primary metastatic disease or within 6 months of last dose of adjuvant therapy
* Presence of at least 1 measurable (target) lesion. Target lesions are defined as those lesions that can be measured in at least 1 dimension as >=20mm with conventional techniques or >=10mm with spiral computerized tomography (CT) scan. Previously irradiated lesions will not be considered as target lesions.
* All previous therapies must have been discontinued at least 4 weeks before study entry, and all acute toxic effects (excluding alopecia or neurotoxicity) of any prior therapy must have resolved to NCI CTC (Version 2.0) Grade <=1 (please see inclusion criteria #8 below for exceptions)
* Age >= 18 years
* ECOG performance status of 0, 1 or 2
* Baseline tests within the following limits: Absolute neutrophil count (ANC) >= 1500/mm3 (1.5 x 10(9)/L) Platelets >= 100,000/mm3 (100 x 10(9)/L) Hemoglobin >= 9.0 g/dL Serum creatinine <= 1.5 mg/dl (or <= 133 mmol/L) Total serum bilirubin <= 1.5 x upper limits of normal (ULN) regardless of liver involvement secondary to tumor SGOT <= 2.5 x ULN; <=5 x ULN if there is liver involvement secondary to tumor Albumin >=3.0 g/dL Pregnancy test for females of childbearing potential is negative within 7 days of starting treatment
* Evidence of personally signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Prior treatment with another topoisomerase I inhibitor
* More than 1 prior chemotherapy regimen for advanced disease
* Prior radiation therapy to >25% of the bone marrow
* Any investigational agent received in the 4 weeks before enrollment to this study and/or current enrollment in another therapeutic clinical trial
* Previous high-dose chemotherapy requiring hematopoietic stem cell rescue
* Known brain metastases, or spinal cord compression, or carcinomatous meningitis (baseline CT or magnetic resonance imaging (MRI) scan of the brain required only in case of clinical suspicion of central nervous system metastases)
* Previous (within the last 5 years) or current malignancies at other sites, except for adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri
* Active inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhea
* Any of the following in the past 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or other significant thromboembolic event
* Ongoing cardiac dysrhythmias of NCI CTC grade >=2, atrial fibrillation of any grade
* Active infection, including known human immunodeficiency virus (HIV) positivity
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. Fertile patients who are refusing to use reliable contraceptive methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To assess the antitumor activity of edotecarin by repeating radiographic assessments at 6-week intervals for all patients.

SECONDARY OUTCOMES:
To determine the time of onset and duration of tumor control, and overall survival.
In addition, the safety and tolerability profile of edotecarin will be assessed, and plasma pharmacokinetic (PK) profile of edotecarin will be evaluated.
Blood samples for PK evaluation will be collected during Cycles 1 and 2 and limited to the patients included in the first stage of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Belgium (3):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, Lille, France
- Spain (2):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Taiwan (2):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Kwei-Shan
- Pfizer Investigational Site, Birmingham, United Kingdom
- Pfizer Investigational Site